CLINICAL TRIAL: NCT02523118
Title: A Prospective, Multicenter Study to Compare and Validate Endoscopic, Histologic, Molecular, and Patient-Reported Outcomes in Pediatric and Adult Patients With Eosinophilic Esophagitis (EoE), Gastritis (EoG), Enteritis (EoN) and Colitis (EoC)
Brief Title: OMEGA: Outcome Measures in Eosinophilic Gastrointestinal Disorders Across the Ages
Acronym: OMEGA
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); ORDR (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-2311; U54AI117870 (Other Grant/Funding Number: NIDDK)
Record Dates: First submitted 2015-06-22; First posted 2015-08-14 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Eosinophilic Gastrointestinal Disorders (EGIDs); Eosinophilic Esophagitis; Eosinophilic Gastritis; Eosinophilic Gastroenteritis; Eosinophilic Colitis
MeSH Terms: conditions — Eosinophilic Esophagitis; Eosinophilic enteropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Biopsies from the gastrointestinal (GI) tract may be collected and used to learn more about eosinophilic gastrointestinal disorders. Genetic analysis may be performed on some of these samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to find the best measures to define how well a person with eosinophilic disorder is doing. People with EoE, EoG, EoN and EoC normally undergo endoscopy and/or colonoscopy where cells are collected for microscopic analysis. Treatments are then decided based on how the cells look. We are aiming to compare different tissue components such as inflammatory cell types with clinical symptoms. We want to see if scores on standard questionnaires can give us an idea how well the person is doing.

DETAILED DESCRIPTION:
This is a longitudinal observational study in which individuals (males and females 3 years of age and greater) with EoE, EoG, EoN and EoC will be followed over the course of time to see if standard questionnaires can give us an idea of how well the person is doing.

Participants undergoing standard of care (normal, routine care) endoscopies and/or colonoscopies will have biopsies (small pieces of tissue from the GI tract normally collected during these procedures) collected and used for the research study. Participants will also complete questionnaires related to their symptoms and quality of life. Participants will be followed over the course of time and asked to complete the questionnaires at various time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 3 years of age and older
* Mucosal eosinophilia:

EoE ≥ 15 eosinophils/HPF in the distal or proximal esophagus EoG ≥ 30 eosinophils/HPF in 5 HPF's in the body and/or antrum EoN ≥ 53 eosinophils/HPF in the duodenum and/or ≥ 56 eosinophils/HPF in the jejunum and/or ileum EoC ≥ 84 eosinophils/HPF from the transverse or descending colon and/or ≥ 32 eosinophils/HPF from the rectosigmoid colon or a biopsy from any colonic location with ≥ 100 eosinophils/HPF

- Presence of symptoms is required for patients who are newly diagnosed but not required for patients who were previously diagnosed.

Exclusion Criteria:

* History of intestinal surgery other than G tube placement
* Enrolled in a blinded investigational study at the time of the first study visit
* Have esophageal stricture (<3mm)
* Have other identifiable causes for eosinophilia (except Inflammatory Bowel Disease): infections, Gastrointestinal (GI) cancer, other GI inflammatory disease (e.g., Ulcerative Colitis or Crohn's Disease)

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females ages 3 or greater with EoE, EoG, EoN or EoC.
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2015-07-17 (Actual); Primary Completion 2050-12-01 (Estimated); Study Completion 2051-01-01 (Estimated)

PRIMARY OUTCOMES:
Mucosal eosinophilia (eos/hpf) | Duration of funding, at least 10 years
  Mucosal eosinophil levels are measured as eosinophils per high power field (eos/hpf). The primary outcome measure is to determine the change in mucosal eosinophil level (eos/hpf) and to determine if the change in mucosal eosinophil level in eos/hpf correlates with the change in scores on clinical outcome measure metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Rothenberg, MD, PhD, Principal Investigator — Cincinnati Children's Hospital Medical Center
Locations (19):
- United States (19):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Arkansas Children's Research Institute, Rogers, Arkansas
  - Rady Children's Hospital, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - Children's Hospital Colorado, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - National Institutes of Health (NIH), Bethesda, Maryland
  - Tufts University, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine & Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Safroneeva E, Pan Z, King E, Martin LJ, Collins MH, Yang GY, Capocelli KE, Arva NC, Abonia JP, Atkins D, Bonis PA, Dellon ES, Falk GW, Gonsalves N, Gupta SK, Hirano I, Leung J, Menard-Katcher PA, Mukkada VA, Schoepfer AM, Spergel JM, Wershil BK, Rothenberg ME, Aceves SS, Furuta GT; Consortium of Eosinophilic Gastrointestinal Disease Researchers. Long-Lasting Dissociation of Esophageal Eosinophilia and Symptoms After Dilation in Adults With Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2022 Apr;20(4):766-775.e4. doi: 10.1016/j.cgh.2021.05.049. Epub 2021 May 29. PMID 34062314
- See also: Learn more about CEGIR at this website. — https://www.rarediseasesnetwork.org/cms/CEGIR